CLINICAL TRIAL: NCT03334903
Title: Gabapentin Regimens and Their Effects on Opioid Consumption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Wolfgang Fitz, M.D., Associate Orthopedic Surgeon, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OpioidNeurontinTKR
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Opioid Use; Opioid Dependence
Keywords: Total Knee Arthroplasty; Neurontin; Gabapentin; Opioid Tapering
MeSH Terms: conditions — Osteoarthritis, Knee; Opioid-Related Disorders | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Standard of care includes one dose of 600 mg gabapentin in the immediate preoperative period (1-2 hours before surgery), then a dose of 600 mg each morning during postoperative admission.
- Postoperative Gabapentin Regimen (Experimental): Single preoperative dose of 600 mg, as described above, plus an additional postoperative regimen. Patients will take 300 mg gabapentin every 8 hours for 1 week after discharge, then a single nightly dose of 300 mg gabapentin for another month.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 600 mg gabapentin before and after surgery. 300 mg gabapentin for approx. 5 weeks after surgery.
  Other Names: Neurontin
  Arms: Postoperative Gabapentin Regimen

SUMMARY:
The purpose of this study is to determine the best strategy of administering gabapentin in connection with our current approach to perioperative pain management. We aim to evaluate two different adjunct gabapentin regimens given in the perioperative period, and to identify which manages patient pain more effectively and safely. In this evaluation, we will identify the quantity of patients' opioid consumption, the quality of their pain management, and the frequency and severity of any side effects they might experience.

Patients who are undergoing total knee replacement (TKR) and choose to participate will be randomly assigned to a treatment group using computer-generated randomization. Patients in group 1 (the control group) will receive the standard of care as pertains to gabapentin. This consists of a single 600 mg dose of gabapentin administered to the patient approximately one to two hours before surgery, then a dose of 600 mg each morning during postoperative admission. Patients in Group 2 will receive 600 mg preoperatively, plus an additional postoperative gabapentin regimen: they will take 300 mg of gabapentin every 8 hours for 1 week, then a single nightly dose of 300 mg for another month.

DETAILED DESCRIPTION:
The purpose of this study is to determine the best strategy of administering gabapentin in connection with our current approach to perioperative pain management. We aim to evaluate two different adjunct gabapentin regimens given in the perioperative period, and to identify which manages patient pain more effectively and safely. In this evaluation, we will identify the quantity of patients' opioid consumption, the quality of their pain management, and the frequency and severity of any side effects they might experience. The target enrollment is 68.

Patients who are undergoing total knee replacement (TKR) at Brigham and Women's Hospital will be informed about the study and asked whether they would like to participate. Upon agreement, a patient will sign his/her consent and will be assigned to a treatment group. Patients in group 1 (the control group) will receive the standard of care as pertains to gabapentin. This consists of a single 600 mg dose of gabapentin administered to the patient approximately one to two hours before surgery, then a dose of 600 mg each morning during postoperative admission. Patients in Group 2 will receive 600 mg preoperatively, plus an additional postoperative gabapentin regimen: they will take 300 mg of gabapentin every 8 hours for 1 week, then a single nightly dose of 300 mg for another month.

Every patient being discharged from the hospital will receive from the nursing staff verbal and written instructions - the latter of which will be either printed or in electronic form - about narcotic medications. The instructions will explain when to use such medications and how to taper off their consumption. Following discharge, patients will take gabapentin as directed by their discharge instructions, and in the process track their opioid consumption on their own in their diaries. They will also document their pain, nausea and satisfaction levels according to the visual analogue scale (VAS). At the first post-operative appointment, patients' levels of opioid use will be verified and compared to the amount recorded in each diary; the actual number of tablets consumed will be compared with the documented amounts and with the prescriptions they received. Patients receiving a new prescription will also receive a matching diary for the total length of opioid treatment, including further directions on how to wean themselves off their medications. Outcome measures will be collected at both post-operative visits, the first occurring 8-10 days after surgery and the second 2-3 months following. Additional data including length of stay, postoperative complications including infection and readmission, Emergency Department visits, and routinely collected postoperative functional outcome measures (PROMs) will be recorded.

The Principal Investigator (PI) will review all drug consumption data and patient-reported outcome measures with the research assistant (RA) on a monthly basis as it is collected. The PI will participate in the collection of outcome data at the first and second postoperative visits. Data which could indicate a potential complication, whether related to the study or not - such as heightened risk of adverse outcomes or non-compliance with the tracking diary - will be addressed by the PI immediately. The PI will determine if the study should be altered in any way or stopped for safety reasons. Reasons for stoppage include a rate of adverse events greater than 10% in either group. Adverse events of primary concern include:

* Excessive sleepiness
* Allergic reactions to the opioid medications or gabapentin

All adverse events are recorded in an adverse event log, which will be kept by the RA throughout the study. The PI will review the data on a monthly basis, as well as whenever the RA alerts the PI to any potential adverse event. These checks will help to ensure validity and patient safety. Unanticipated problems will be reported to the PHRC in accordance with PHRC guidelines.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Receiving surgery for total knee replacement (TKR)
* Opioid naïve
* Agrees to use tracking diary to monitor opioid consumption

Exclusion Criteria:

* Over 75 years of age on the date of surgery
* If female, pregnant
* Has received investigational articles < 30 days prior to enrollment or is currently receiving investigational products or devices
* Chronic pain syndrome
* Taking chronic narcotics and/or taking more than 10 mg of codeine per day, any amount of Hydrocodone, over 200 mg of tramadol per day, or any other narcotics prescribed for moderate or severe pain
* Involved in pain clinics for chronic pain, or pain that is not related to the surgical site
* On long-term gabapentin regimen
* Taking Lyrica or Gralise
* Known history of depression or has been treated for depression with medication
* Has entertained suicidal thoughts and behaviors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fitz, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bannister K, Qu C, Navratilova E, Oyarzo J, Xie JY, King T, Dickenson AH, Porreca F. Multiple sites and actions of gabapentin-induced relief of ongoing experimental neuropathic pain. Pain. 2017 Dec;158(12):2386-2395. doi: 10.1097/j.pain.0000000000001040. PMID 28832395
- [Background] Ozgencil E, Yalcin S, Tuna H, Yorukoglu D, Kecik Y. Perioperative administration of gabapentin 1,200 mg day-1 and pregabalin 300 mg day-1 for pain following lumbar laminectomy and discectomy: a randomised, double-blinded, placebo-controlled study. Singapore Med J. 2011 Dec;52(12):883-9. PMID 22159931
- [Background] Rusy LM, Hainsworth KR, Nelson TJ, Czarnecki ML, Tassone JC, Thometz JG, Lyon RM, Berens RJ, Weisman SJ. Gabapentin use in pediatric spinal fusion patients: a randomized, double-blind, controlled trial. Anesth Analg. 2010 May 1;110(5):1393-8. doi: 10.1213/ANE.0b013e3181d41dc2. PMID 20418301
- [Background] Stock CJ, Carpenter L, Ying J, Greene T. Gabapentin versus chlordiazepoxide for outpatient alcohol detoxification treatment. Ann Pharmacother. 2013 Jul-Aug;47(7-8):961-9. doi: 10.1345/aph.1R751. Epub 2013 Jun 18. PMID 23780805
- [Background] Mason BJ, Quello S, Goodell V, Shadan F, Kyle M, Begovic A. Gabapentin treatment for alcohol dependence: a randomized clinical trial. JAMA Intern Med. 2014 Jan;174(1):70-7. doi: 10.1001/jamainternmed.2013.11950. PMID 24190578
- [Background] Leung JG, Hall-Flavin D, Nelson S, Schmidt KA, Schak KM. The role of gabapentin in the management of alcohol withdrawal and dependence. Ann Pharmacother. 2015 Aug;49(8):897-906. doi: 10.1177/1060028015585849. Epub 2015 May 12. PMID 25969570
- [Background] Grant MC, Lee H, Page AJ, Hobson D, Wick E, Wu CL. The Effect of Preoperative Gabapentin on Postoperative Nausea and Vomiting: A Meta-Analysis. Anesth Analg. 2016 Apr;122(4):976-85. doi: 10.1213/ANE.0000000000001120. PMID 26991615
- [Background] Misra S, Parthasarathi G, Vilanilam GC. The effect of gabapentin premedication on postoperative nausea, vomiting, and pain in patients on preoperative dexamethasone undergoing craniotomy for intracranial tumors. J Neurosurg Anesthesiol. 2013 Oct;25(4):386-91. doi: 10.1097/ANA.0b013e31829327eb. PMID 23603887
- [Background] Montazeri K, Kashefi P, Honarmand A. Pre-emptive gabapentin significantly reduces postoperative pain and morphine demand following lower extremity orthopaedic surgery. Singapore Med J. 2007 Aug;48(8):748-51. PMID 17657384
- [Background] Rai AS, Khan JS, Dhaliwal J, Busse JW, Choi S, Devereaux PJ, Clarke H. Preoperative pregabalin or gabapentin for acute and chronic postoperative pain among patients undergoing breast cancer surgery: A systematic review and meta-analysis of randomized controlled trials. J Plast Reconstr Aesthet Surg. 2017 Oct;70(10):1317-1328. doi: 10.1016/j.bjps.2017.05.054. Epub 2017 Jun 9. PMID 28751024
- [Background] Arumugam S, Lau CS, Chamberlain RS. Use of preoperative gabapentin significantly reduces postoperative opioid consumption: a meta-analysis. J Pain Res. 2016 Sep 12;9:631-40. doi: 10.2147/JPR.S112626. eCollection 2016. PMID 27672340
- [Background] Hassani V, Pazouki A, Nikoubakht N, Chaichian S, Sayarifard A, Shakib Khankandi A. The effect of gabapentin on reducing pain after laparoscopic gastric bypass surgery in patients with morbid obesity: a randomized clinical trial. Anesth Pain Med. 2015 Feb 1;5(1):e22372. doi: 10.5812/aapm.22372. eCollection 2015 Feb. PMID 25789237
- [Background] Mardani-Kivi M, Mobarakeh MK, Keyhani S, Motlagh KH, Ekhtiari KS. Is gabapentin effective on pain management after arthroscopic anterior cruciate ligament reconstruction? A triple blinded randomized controlled trial. Arch Bone Jt Surg. 2013 Sep;1(1):18-22. Epub 2013 Sep 15. PMID 25207278
- [Background] Chiu TW, Leung CC, Lau EY, Burd A. Analgesic effects of preoperative gabapentin after tongue reconstruction with the anterolateral thigh flap. Hong Kong Med J. 2012 Feb;18(1):30-4. PMID 22302908
- [Background] Moore A, Costello J, Wieczorek P, Shah V, Taddio A, Carvalho JC. Gabapentin improves postcesarean delivery pain management: a randomized, placebo-controlled trial. Anesth Analg. 2011 Jan;112(1):167-73. doi: 10.1213/ANE.0b013e3181fdf5ee. Epub 2010 Nov 16. PMID 21081764
- [Background] Menda F, Koner O, Sayin M, Ergenoglu M, Kucukaksu S, Aykac B. Effects of single-dose gabapentin on postoperative pain and morphine consumption after cardiac surgery. J Cardiothorac Vasc Anesth. 2010 Oct;24(5):808-13. doi: 10.1053/j.jvca.2009.10.023. Epub 2010 Jan 6. PMID 20056448
- [Background] Ture H, Sayin M, Karlikaya G, Bingol CA, Aykac B, Ture U. The analgesic effect of gabapentin as a prophylactic anticonvulsant drug on postcraniotomy pain: a prospective randomized study. Anesth Analg. 2009 Nov;109(5):1625-31. doi: 10.1213/ane.0b013e3181b0f18b. Epub 2009 Aug 27. PMID 19713257
- [Background] Clivatti J, Sakata RK, Issy AM. Review of the use of gabapentin in the control of postoperative pain. Rev Bras Anestesiol. 2009 Jan-Feb;59(1):87-98. doi: 10.1590/s0034-70942009000100012. English, Portuguese. PMID 19374220
- [Background] Pandey CK, Navkar DV, Giri PJ, Raza M, Behari S, Singh RB, Singh U, Singh PK. Evaluation of the optimal preemptive dose of gabapentin for postoperative pain relief after lumbar diskectomy: a randomized, double-blind, placebo-controlled study. J Neurosurg Anesthesiol. 2005 Apr;17(2):65-8. doi: 10.1097/01.ana.0000151407.62650.51. PMID 15840990
- [Background] Dierking G, Duedahl TH, Rasmussen ML, Fomsgaard JS, Moiniche S, Romsing J, Dahl JB. Effects of gabapentin on postoperative morphine consumption and pain after abdominal hysterectomy: a randomized, double-blind trial. Acta Anaesthesiol Scand. 2004 Mar;48(3):322-7. doi: 10.1111/j.0001-5172.2004.0329.x. PMID 14982565
- [Background] Ho KY, Gan TJ, Habib AS. Gabapentin and postoperative pain--a systematic review of randomized controlled trials. Pain. 2006 Dec 15;126(1-3):91-101. doi: 10.1016/j.pain.2006.06.018. Epub 2006 Jul 18. PMID 16846695
- [Background] Ucak A, Onan B, Sen H, Selcuk I, Turan A, Yilmaz AT. The effects of gabapentin on acute and chronic postoperative pain after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Oct;25(5):824-9. doi: 10.1053/j.jvca.2010.11.017. Epub 2011 Jan 12. PMID 21232979
- [Background] Clarke H, Pereira S, Kennedy D, Gilron I, Katz J, Gollish J, Kay J. Gabapentin decreases morphine consumption and improves functional recovery following total knee arthroplasty. Pain Res Manag. 2009 May-Jun;14(3):217-22. doi: 10.1155/2009/930609. PMID 19547761
- [Background] Smith RV, Havens JR, Walsh SL. Gabapentin misuse, abuse and diversion: a systematic review. Addiction. 2016 Jul;111(7):1160-74. doi: 10.1111/add.13324. Epub 2016 Mar 18. PMID 27265421
- [Background] Menigaux C, Adam F, Guignard B, Sessler DI, Chauvin M. Preoperative gabapentin decreases anxiety and improves early functional recovery from knee surgery. Anesth Analg. 2005 May;100(5):1394-1399. doi: 10.1213/01.ANE.0000152010.74739.B8. PMID 15845693

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Started | 39 | 38
Completed | 35 | 33
Not Completed | 4 | 5
Not completed — Use of medical marijuana - determined ineligible later in study | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Surgery postponed | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 68 total patients completed study, after dropout of 9 total participants from overall number enrolled
  years | 64.6 (6.8) | 64.2 (6.7) | 64.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 17 | 16 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (4.5) | 32.1 (5.3) | 31.2 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Mean opioid consumption, measured in mg of morphine equivalents.
Time Frame: 2-3 months following surgery (total amount measured at second postoperative appointment; means assessed afterwards).
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
morphine equivalents | 287.0 (227.99) | 281.1 (230.31)

2. Secondary Outcome: Days Taking Opioids
Description: Number of days until patients are finished consuming opioid medications after discharge.
Time Frame: 2-3 months following surgery (measured at second postoperative appointment).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
days | 14.8 (10.69) | 18.7 (18.57)

3. Secondary Outcome: VAS Score 1: "How Much Pain do You Feel in Your Operative Site When Resting?"
Description: Surgical site pain. Scale 0-10, with 0 best and 10 worst
Time Frame: 2-3 months after surgery (at 2nd postoperative appointment)
Measure: Mean (Standard Deviation); unit: score on 10-point scale
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
score on 10-point scale | 2.26 (1.36) | 2.46 (1.57)

4. Secondary Outcome: VAS Score 2: "How Much Pain do You Feel in Your Operative Site When Moving?"
Description: Surgical site pain. Scale 0-10, with 0 best and 10 worst.
Time Frame: 2-3 months following surgery (measured at second postoperative appointment).
Measure: Mean (Standard Deviation); unit: score on a 10-point scale
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
score on a 10-point scale | 3.84 (1.54) | 3.54 (1.54)

5. Secondary Outcome: VAS Score 3: "How Well Are You Sleeping?"
Description: Sleep quality. Scale 0-10 with 0 worst and 10 best.
Time Frame: 2-3 months following surgery (measured at second postoperative appointment).
Measure: Mean (Standard Deviation); unit: score on a 10-point scale
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
score on a 10-point scale | 5.73 (2.16) | 6.38 (1.75)

6. Secondary Outcome: VAS Score 4: "How Bad is Your Nausea?"
Description: Nausea. Scale 0-10, with 0 best and 10 worst.
Time Frame: 2-3 months following surgery (measured at second postoperative appointment).
Measure: Mean (Standard Deviation); unit: score on a 10-point scale
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
score on a 10-point scale | 0.36 (0.53) | 0.17 (0.40)

7. Secondary Outcome: VAS Score 5: "How Satisfied Are You With Your Pain Management?"
Description: Satisfaction. Scale 0-10 with 0 worst and 10 best.
Time Frame: 2-3 months following surgery (measured at second postoperative appointment).
Measure: Mean (Standard Deviation); unit: score on a 10-point scale
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
Number analyzed (Participants) | 35 | 33
score on a 10-point scale | 7.83 (2.23) | 8.48 (1.39)

ADVERSE EVENTS:
Time Frame: Adverse events collected through study completion, an average of 3 months
Arm/Group | Standard of Care | Postoperative Gabapentin Regimen
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 1/39 | 1/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=39) | Postoperative Gabapentin Regimen (N=38)
Dizziness (General disorders) | 0 (0) | 1 (1)
GI Distress (Gastrointestinal disorders) | 1 (1) | 0 (0) — GI distress from anesthesia / narcotics post-operative

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03334903/Prot_SAP_000.pdf